CLINICAL TRIAL: NCT05062863
Title: A Prospective, Observational Clinical Study of the Safety, Effectiveness and Clinical Benefits of the T3 Dental Implant System
Brief Title: An Observational Clinical Study of the T3 Dental Implant System
Acronym: Kashmir
Status: Active, not recruiting | Type: Observational
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 1804
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: T3 dental implant system — This clinical study will evaluate patients being treated with the T3 dental implant to confirm its safety and performance (effect of treatment of edentulism). The patients treated will experience a benefit from treatment of edentulism with the T3 dental implant system. The patients will be followed prospectively from the time of exposure (dental implant placement surgery) to outcome (implant survival at 2 years).
  Other Names: T3 platform switched certain parallel walled (BOPS); T3 non-platform switched certain parallel walled (BOSS); T3 with DCD platform switched certain parallel walled (BNPS); T3 with DCD non-platform switched certain parallel walled (BNSS)

SUMMARY:
This will be a prospective, observational study where all implants will be placed in either the maxilla or mandible and loaded immediately (within 48 hours), early (within 6-8 weeks) or delayed (> 8 weeks) with a provisional or definitive prosthesis. The implants will be evaluated yearly for 2 years.

DETAILED DESCRIPTION:
This study aims to enroll a total of 140 patients (140 implants) who are in need of treatment with dental implants in one or more edentulous areas of the maxilla and/or mandible. Approximately 4 sites will be participating, each one contributing 35 patients to the study dataset.

The main objectives of this study will be:

1. The integration success of the dental implant (as measured by mobility)
2. The measured changes in peri-implant crestal bone levels for each implant
3. Confirmation of clinical benefits

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex and at least 18 years of age.
2. Patients for whom a decision has already been made to use a dental implant for the restoration of existing edentulism in the mandible and/or maxilla.
3. Prior extracted sites or simultaneous extraction/implant placement.
4. Patients must be physically able to tolerate conventional surgical and restorative procedures.
5. Patients who provide a signed informed consent.
6. Patients who agree to be evaluated for each study visit.

Exclusion Criteria:

1. Patients who are known to be pregnant at the screening visit or planning to become pregnant within 6 months of study enrollment.
2. Patients who have previously failed dental implants at the site intended for study implant placement.
3. Patients with active HIV or Hepatitis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Qualified patient will be those patients who have been newly diagnosed with needing a dental implant (or more than one) in one or more edentulous areas in the maxilla and/or mandible. Patients who have had prior implants in the treatment site that have failed (in need of revision) are not eligible for inclusion.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Dental implant integration | 2 years
  The integration success measured by lack of mobility

SECONDARY OUTCOMES:
Crestal Bone Loss | 2 years
  The measured changes in peri-implant crestal bone levels

CONTACTS AND LOCATIONS:
Overall Officials: Hai Bo Wen, PhD, Study Director — ZimVie
Locations (4):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Virginia Commonwealth University, Richmond, Virginia
- Dr. Daniel Engler-Hamm, München, Germany

IPD SHARING:
Plan to Share IPD: No